CLINICAL TRIAL: NCT04990076
Title: Ultrasound Evaluation of the Myometrium Using the MUSA Terminology, Comparison With Histology.
Brief Title: Ultrasound Evaluation of the Myometrium Using the MUSA Terminology Comparison With Histology
Acronym: MUSA1
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s62497
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Myoma;Uterus; Sarcoma Uterus
MeSH Terms: conditions — Myofibroma | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients planned for hysterectomy with a myometrial lesion of more than 1 cm.
  Interventions: Procedure: Hysterectomy

INTERVENTIONS:
Procedure: Hysterectomy — Surgery includes different types of hysterectomy: vaginal hysterectomy, total abdominal hysterectomy and laparoscopic or Robotic hysterectomy. The type of hysterectomy does not influence histological outcome, as long as the uterus is removed in one part (no power morcellation). Indications for surgery and the type of surgery are according to the departments' protocols. If the patient is deemed to be inoperable due to the extent of the disease, a representive biopsy (e.g. trucut biopsy) will be accepted if sufficiently motivated by the oncology team.

SUMMARY:
The main objective is to evaluate the diagnostic accuracy of the MUSA terms and definitions, as defined in the paper by Van den Bosch T, Dueholm M, ea. in 2015, to differentiate between different types of myometrial lesions of more than 1 cm. The primary aim is the diagnostic accuracy of the MUSA terms and definitions and the secondary aim the development of a prediction model.

DETAILED DESCRIPTION:
Primary aim: Diagnostic accuracy of the MUSA terms and definitions

Every patient planned for hysterectomy for myometrial pathology (e.g. benign fibroid, benign adenomyoma or malignant uterine sarcoma) will undergo a systematic preoperative ultrasound scan. Around 50 ultrasound characteristics will be assess as to diagnostic accuracy as predictors (Prospective evaluation of MUSA terms and definitions). The estimation for sarcomas is based on preliminary and unpublished results from an ongoing prospective study led by prof dr Antonia Testa from the Università Cattolica di Sacro Cuore Largo Agostino Gemelli in Rome showing an incidence of 4.9% for uterine sarcomas amongst women with a myometrial lesion referred to their tertiary center (Antonia Testa, personal communication).

Secondary aim: Development of prediction model

The Secondary aim is to build predictive models to differentiate between benign myometrial lesions (e.g. adenomyosis and fibroid) and malignant myometrial lesion (e.g. uterine sarcoma). Because of the small number of cases with malignant myometrial lesion (expected to be 5% of the study population or around 75 women), we will limit the number of variables to be tested in order to avoid overfitting. Based on current literature, we preselected following characteristics for development of a prediction model:

* Outer contour: regular of irregular
* Echogenicity of uterine lesion: uniform (homogeneous) or non-uniform (mixed)
* Colour score: 1 to 4
* Presence of central necrosis
* Maximal diameter of the lesion (in mm)
* Presence of acoustic shadows

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients planned to undergo hysterectomy for myometrial pathology of more then 1cm (e.g. fibroid, focal adenomyosis, uterine sarcoma).

Exclusion Criteria:

* Patient's refusal
* Age < 18 years
* Polymyomatous uterus
* Myometrial lesion with a diameter less then 10mm
* Patients currently treated for another cancer
* Patients with ovarian pathology, endometrial pathology of cervical pathology
* Power morcellation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for hysterectomy with a myometrial lesion
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the MUSA terms and definitions | 4 years
  Around 50 ultrasound characteristics will be assess as to diagnostic accuracy as predictors (Prospective evaluation of MUSA terms and definitions).

SECONDARY OUTCOMES:
Development of prediction model | 5 years
  predictive models to differentiate between benign myometrial lesions (e.g. adenomyosis and fibroid) and malignant myometrial lesion (e.g. uterine sarcoma).

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Timmerman, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van den Bosch T, Dueholm M, Leone FP, Valentin L, Rasmussen CK, Votino A, Van Schoubroeck D, Landolfo C, Installe AJ, Guerriero S, Exacoustos C, Gordts S, Benacerraf B, D'Hooghe T, De Moor B, Brolmann H, Goldstein S, Epstein E, Bourne T, Timmerman D. Terms, definitions and measurements to describe sonographic features of myometrium and uterine masses: a consensus opinion from the Morphological Uterus Sonographic Assessment (MUSA) group. Ultrasound Obstet Gynecol. 2015 Sep;46(3):284-98. doi: 10.1002/uog.14806. Epub 2015 Aug 10. PMID 25652685
- [Background] Ludovisi M, Moro F, Pasciuto T, Di Noi S, Giunchi S, Savelli L, Pascual MA, Sladkevicius P, Alcazar JL, Franchi D, Mancari R, Moruzzi MC, Jurkovic D, Chiappa V, Guerriero S, Exacoustos C, Epstein E, Fruhauf F, Fischerova D, Fruscio R, Ciccarone F, Zannoni GF, Scambia G, Valentin L, Testa AC. Imaging in gynecological disease (15): clinical and ultrasound characteristics of uterine sarcoma. Ultrasound Obstet Gynecol. 2019 Nov;54(5):676-687. doi: 10.1002/uog.20270. Epub 2019 Oct 7. PMID 30908820